CLINICAL TRIAL: NCT03165877
Title: Effect of Low-glycemic Index Lunches and Dinners Intake on Indicators of Satiety, Metabolic Parameters and Liver Steatosis Degree on Women With Type 2 Diabetes Under Metformin Therapy: Controlled Clinical Trial
Brief Title: Effect of Low-glycemic Index Meals Intake on DM2 Women Under Metformin Therapy
Acronym: LGIM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Valparaiso (Other)
Responsible Party: Principal Investigator, Claudia Vega Soto, Nutritionist, Universidad de Valparaiso
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 035-2013
Record Dates: First submitted 2017-05-20; First posted 2017-05-24 (Actual); Last update posted 2017-05-24 (Actual); Status verified 2017-05

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: GLYCEMIC INDEX; NAFLD; METABOLIC PARAMETERS; SATIETY
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Low-glycemic index (Experimental): Low-glycemic index lunches and dinners (<55%)
  Interventions: Other: Low-glycemic index
- Control (Active Comparator): Medium/high glycemic index lunches and dinners (>60%)
  Interventions: Other: Control

INTERVENTIONS:
Other: Low-glycemic index — Subjects ate low-glycemic index lunches and dinners (<55%),consisting of salad, main course and dessert, respectively.
  Arms: Low-glycemic index
Other: Control — Subjects ate standard lunches and dinners (>60%),consisting of salad, main course and dessert, respectively.
  Arms: Control

SUMMARY:
To compare the effect of low-glycemic index versus control lunches and dinners intake on indicators of satiety, metabolic parameters and liver steatosis degree on women with type 2 diabetes under metformin therapy.

ELIGIBILITY:
Inclusion Criteria:

* Subjets with type 2 diabetes mellitus diagnosis under metformin therapy.
* Female sex.
* Aged 30 to 65 years.
* Body Mass Index (BMI) 22 to 34.9 kg / m2.

Exclusion Criteria:

* Women with insulin-releasing drugs or insulin treatment.
* Patients with diabetic nephropathy, retinopathy, chronic kidney disease, stroke.
* Subjects with hypothyroidism without treatment.
* Individuals with food allergies or intolerances.
* Women who present an intake of ≥20 g of alcohol per day quantified through a closed consumption frequency survey.
* Patients with previously diagnosed hepatitis, hepatic cirrhosis or liver cancer.

Ages: 30 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2016-05-31 (Actual); Primary Completion 2016-10-13 (Actual); Study Completion 2016-10-13 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Fasting glycemia at 12 weeks | up to 12 weeks
  Fasting glycemia (mg/dL) was measured at Baseline and at 12 weeks
Postprandial glycemia | up to 12 weeks
  Postprandial glycemia (mg/dL) was measured for lunch and dinner of one day at 4, 8 and 12 weeks
Change from Baseline Glycosylated hemoglobin at 12 weeks | up to 12 weeks
  Glycosylated hemoglobin was measured at Baseline and at 12 weeks
Change from Baseline Triglycerides at 12 weeks | up to 12 weeks
  Triglycerides (mg/dL) was measured at Baseline and at 12 weeks
Change from Baseline Total cholesterol/HDL ratio at 12 weeks | up to 12 weeks
  Total cholesterol/HDL ratio was measured at Baseline and at 12 weeks
Change from Baseline HDL cholesterol at 12 weeks | up to 12 weeks
  HDL cholesterol (mg/dL) was measured at Baseline and at 12 weeks
Change from Baseline Total cholesterol at 12 weeks | up to 12 weeks
  Total cholesterol (mg/dL) was measured at Baseline and at 12 weeks
Change from Baseline LDL cholesterol at 12 weeks | up to 12 weeks
  LDL cholesterol (mg/dL) was measured at Baseline and at 12 weeks
Change from Baseline High-sensitivity C-reactive protein (hs-CRP) at 12 weeks | up to 12 weeks
  High-sensitivity C-reactive protein (mg/L) was measured at Baseline and at 12 weeks
Change from Baseline Aspartate aminotransferase (AST) at 12 weeks | up to 12 weeks
  Aspartate aminotransferase (UI/L) was measured at Baseline and at 12 weeks
Change from Baseline Alanine aminotransferase (ALT) at 12 weeks | up to 12 weeks
  Alanine aminotransferase (UI/L) was measured at Baseline and at 12 weeks
Change from Baseline Liver steatosis degree at 12 weeks | up to 12 weeks
  Liver steatosis degree was measured at Baseline, 4, 8 and 12 weeks
Subjective satiety | 7 days
  Visual Analog Scale (VAS) was applied after lunches and dinners of 7 days to each subject
Objective satiety | 7 days
  24-hour recall was applied the same 7 days as the VAS to each subject

SECONDARY OUTCOMES:
Body mass index (BMI) | up to 12 weeks
  Body mass index (BMI) (kg/m2) was measured at Baseline, 4, 8 and 12 weeks.
Waist circumference | up to 12 weeks
  Waist circumference (cm) was measured at Baseline, 4, 8 and 12 weeks.
Alcohol intake | up to 12 weeks
  Alcohol intake (g/day) was measured at Baseline, 4, 8 and 12 weeks.
Physical activity | up to 12 weeks
  Physical activity was measured at Baseline, 4, 8 and 12 weeks.
Adherence to treatment | up to 12 weeks
  The percentage of adherence to treatment was measured through a daily survey for 12 weeks. It is the calculation of compliance with planned meals intake (number of lunches and dinners eaten / total number of lunches and dinners of the study x 100).

IPD SHARING:
Plan to Share IPD: No